CLINICAL TRIAL: NCT04407117
Title: Change in the Incidence of Appendicitis in a Controlled Environment During the National Lockdown Throughout the COVID-19 Pandemic
Brief Title: Appendicitis During the National Lockdown During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Claus Anders Bertelsen, PhD, MD (Other)
Responsible Party: Sponsor-Investigator, Claus Anders Bertelsen, PhD, MD, Associate professor, consultant surgeon, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Other Study IDs: APPCOVID-19
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-06-19 (Actual); Status verified 2020-06

CONDITIONS: Appendicitis
Keywords: COVID-19; Pandemic; Incidence
MeSH Terms: conditions — Appendicitis; COVID-19 | interventions — Physical Distancing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Lock-down and social distancing — Lock-down and social distancing during COVID-19 pandemic

SUMMARY:
The study aims to examine whether a nationwide lock-down with an entire population subjugated to social distancing reduces the incidence of appendicitis. If a reduction is detected it supports the hypothesis that infectious disease may play a role in the etiology of appendicitis.

ELIGIBILITY:
Inclusion Criteria:

Registered in the Danish National Patient Register during the study period

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All persons registered in the Danish National Patient Register, i.e. all persons resident in Denmark
Sampling Method: Non-Probability Sample
Enrollment: 6000000 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2020-04-19 (Actual); Study Completion 2020-04-19 (Actual)

PRIMARY OUTCOMES:
Appendectomy | 5 weeks
  Appendectomy or other surgery for appendicitis

SECONDARY OUTCOMES:
Postoperative length of stay | 30 days
  Postoperative length of stay
Mortality | 30 days
  Overall mortality
Incidence of complicated appendicitis | 5 weeks
  Perforated appendicitis or periappendicular abscess

CONTACTS AND LOCATIONS:
Overall Officials: Claus A Bertelsen, PhD, Study Director — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Addiss DG, Shaffer N, Fowler BS, Tauxe RV. The epidemiology of appendicitis and appendectomy in the United States. Am J Epidemiol. 1990 Nov;132(5):910-25. doi: 10.1093/oxfordjournals.aje.a115734. PMID 2239906
- [Background] Bhangu A, Soreide K, Di Saverio S, Assarsson JH, Drake FT. Acute appendicitis: modern understanding of pathogenesis, diagnosis, and management. Lancet. 2015 Sep 26;386(10000):1278-1287. doi: 10.1016/S0140-6736(15)00275-5. PMID 26460662
- [Background] Lamps LW. Infectious causes of appendicitis. Infect Dis Clin North Am. 2010 Dec;24(4):995-1018, ix-x. doi: 10.1016/j.idc.2010.07.012. PMID 20937462
- [Background] Dzabic M, Bostrom L, Rahbar A. High prevalence of an active cytomegalovirus infection in the appendix of immunocompetent patients with acute appendicitis. Inflamm Bowel Dis. 2008 Feb;14(2):236-41. doi: 10.1002/ibd.20299. PMID 17973298
- [Background] Carr NJ. The pathology of acute appendicitis. Ann Diagn Pathol. 2000 Feb;4(1):46-58. doi: 10.1016/s1092-9134(00)90011-x. PMID 10684382
- [Background] Hsu YJ, Fu YW, Chin T. Seasonal variations in the occurrence of acute appendicitis and their relationship with the presence of fecaliths in children. BMC Pediatr. 2019 Nov 16;19(1):443. doi: 10.1186/s12887-019-1824-9. PMID 31731890
- [Background] Wei PL, Chen CS, Keller JJ, Lin HC. Monthly variation in acute appendicitis incidence: a 10-year nationwide population-based study. J Surg Res. 2012 Dec;178(2):670-6. doi: 10.1016/j.jss.2012.06.034. Epub 2012 Jul 6. PMID 22795352
- [Background] Stein GY, Rath-Wolfson L, Zeidman A, Atar E, Marcus O, Joubran S, Ram E. Sex differences in the epidemiology, seasonal variation, and trends in the management of patients with acute appendicitis. Langenbecks Arch Surg. 2012 Oct;397(7):1087-92. doi: 10.1007/s00423-012-0958-0. Epub 2012 Jun 2. PMID 22661078
- [Background] Ilves I, Fagerstrom A, Herzig KH, Juvonen P, Miettinen P, Paajanen H. Seasonal variations of acute appendicitis and nonspecific abdominal pain in Finland. World J Gastroenterol. 2014 Apr 14;20(14):4037-42. doi: 10.3748/wjg.v20.i14.4037. PMID 24833844
- [Background] Reinisch A, Heil J, Woeste G, Bechstein W, Liese J. The meteorological influence on seasonal alterations in the course of acute appendicitis. J Surg Res. 2017 Sep;217:137-143. doi: 10.1016/j.jss.2017.05.015. Epub 2017 May 10. PMID 28599958
- [Background] Lynge E, Sandegaard JL, Rebolj M. The Danish National Patient Register. Scand J Public Health. 2011 Jul;39(7 Suppl):30-3. doi: 10.1177/1403494811401482. PMID 21775347
- [Background] Pedersen CB. The Danish Civil Registration System. Scand J Public Health. 2011 Jul;39(7 Suppl):22-5. doi: 10.1177/1403494810387965. PMID 21775345
- [Background] Kleif J, Thygesen LC, Gogenur I. Validity of the diagnosis of appendicitis in the Danish National Patient Register. Scand J Public Health. 2020 Feb;48(1):38-42. doi: 10.1177/1403494818761765. Epub 2018 Mar 19. PMID 29554842
- [Derived] Jantzen AT, Bang-Nielsen A, Bertelsen CA, Torp-Pedersen C, Kleif J. Incidence of appendicitis during COVID-19 lockdown: A nationwide population-based study. Scand J Surg. 2022 Apr-Jun;111(2):14574969221089387. doi: 10.1177/14574969221089387. PMID 35488422